CLINICAL TRIAL: NCT01535638
Title: Relative Bioavailability of BI 207127 FF Tablets, BI 207127 FF Modified Tablets and BI 207127 TFII Tablets Administered Orally as Three Tablets (Single Dose) to Healthy Male Volunteers, an Open-label, Randomised Three-way Crossover Study
Brief Title: Bioavailability of 3 Different Formulations of BI 207127 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1241.26
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — deleobuvir

ARMS (3):
- BI 207127 NA TFII medium dose (Active Comparator): Film-coated tablet for oral administration
  Interventions: Drug: BI 207127
- BI 207127 NA FF medium dose (Active Comparator): Film-coated tablet for oral administration
  Interventions: Drug: BI 207127
- BI 207127 NA FF modified medium dose (Active Comparator): Film-coated tablet for oral administration
  Interventions: Drug: BI 207127

INTERVENTIONS:
Drug: BI 207127 — Medium dose film-coated tablet
  Arms: BI 207127 NA FF modified medium dose
Drug: BI 207127 — Medium dose film-coated tablet
  Arms: BI 207127 NA FF medium dose
Drug: BI 207127 — Medium dose film-coated tablet
  Arms: BI 207127 NA TFII medium dose

SUMMARY:
The primary objective of the current study is to investigate the relative bioavailability of three trial formulations of BI 207127, the trial formulation 2 (TFII), the final formulation (FF), and a FF modified formulation. All formulations are supplied as film-coated Tablets and administered as single dose treatments of BI 207127 (3 film-coated Tablets) in healthy volunteers, with the aim to compare the bioavailability of the three formulations. All treatments will be applied fed, 30 minutes after start of the intake of a standard normal breakfast.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to a complete medical history, including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age =21and Age =50 years
3. Body mass index =18.5 and BMI = 29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least 10 half-lifes prior to administration of the trial drug or during the trial
10. Use of drugs which might reasonably influence the results of the trial within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration of the trial drug or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Alcohol abuse (more than 40 g/day)
14. Drug abuse
15. Blood donation (more than 100 mL within four weeks prior to first administration of the trial drug or during the trial)
16. Excessive physical activities (within one week prior to first administration of the trial drug or during the trial)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of trial site
19. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
20. A history of additional risk factors for Torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
21. History of photosensitivity or recurrent rash
22. Subject is not willing to avoid sun exposure from the first administration of the trial drug until the end of the study.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.26.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Trial Formulation II / Final Formulation (FF) / FF Modified: In this sequence group the treatments (600 mg Deleobuvir in different formulations, single dose) are administered in the order Trial Formulation (TF) II, Final Formulation (FF) and FF modified. There was a wash out period of at least 6 days between each drug administration.
- Trial Formulation II / Final Formulation (FF) Modified / FF: In this sequence group the treatments (600 mg Deleobuvir in different formulations, single dose) are administered in the order Trial Formulation II, Final Formulation modified and Final Formulation. There was a wash out period of at least 6 days between each drug administration.
- Final Formulation (FF) / Trial Formulation II / FF Modified: In this sequence group the treatments (600 mg Deleobuvir in different formulations, single dose) are administered in the order Final Formulation, Trial Formulation II and Final Formulation modified. There was a wash out period of at least 6 days between each drug administration.
- Final Formulation (FF) / FF Modified / Trial Formulation II: In this sequence group the treatments (600 mg Deleobuvir in different formulations, single dose) are administered in the order Final Formulation, Final Formulation modified and Trial Formulation II. There was a wash out period of at least 6 days between each drug administration.
- Final Formulation (FF) Modified / Trial Formulation II / FF: In this sequence group the treatments (600 mg Deleobuvir in different formulations, single dose) are administered in the order Final Formulation modified, Trial Formulation II and Final Formulation. There was a wash out period of at least 6 days between each drug administration.
- Final Formulation (FF) Modified / FF / Trial Formulation II: In this sequence group the treatments (600 mg Deleobuvir in different formulations, single dose) are administered in the order Final Formulation modified, Final Formulation and Trial Formulation II. There was a wash out period of at least 6 days between each drug administration.
Period: Treatment 1 (Single Dose)
Arm/Group | Trial Formulation II / Final Formulation (FF) / FF Modified | Trial Formulation II / Final Formulation (FF) Modified / FF | Final Formulation (FF) / Trial Formulation II / FF Modified | Final Formulation (FF) / FF Modified / Trial Formulation II | Final Formulation (FF) Modified / Trial Formulation II / FF | Final Formulation (FF) Modified / FF / Trial Formulation II
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment 2 (Single Dose)
Arm/Group | Trial Formulation II / Final Formulation (FF) / FF Modified | Trial Formulation II / Final Formulation (FF) Modified / FF | Final Formulation (FF) / Trial Formulation II / FF Modified | Final Formulation (FF) / FF Modified / Trial Formulation II | Final Formulation (FF) Modified / Trial Formulation II / FF | Final Formulation (FF) Modified / FF / Trial Formulation II
Started | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 3 (Single Dose)
Arm/Group | Trial Formulation II / Final Formulation (FF) / FF Modified | Trial Formulation II / Final Formulation (FF) Modified / FF | Final Formulation (FF) / Trial Formulation II / FF Modified | Final Formulation (FF) / FF Modified / Trial Formulation II | Final Formulation (FF) Modified / Trial Formulation II / FF | Final Formulation (FF) Modified / FF / Trial Formulation II
Started | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 3 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: This study was conducted in healthy male subjects as open-label, single-dose, randomised three-way crossover trial to investigate relative bioavailability. Each subject was planned to receive all 3 treatments in a randomly assigned order. The treatments were 3 single doses of 600 mg (3 film-coated tablets à 200 mg each) of Deleobuvir, either as TF II (trial formulation 2) formulation, FF (final formulation) formulation or as FF modified formulation.
Arm/Group | All Subjects
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: AUC0-∞
Description: Area under the concentration-time curve of Deleobuvir in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: 1:00 (h) hour before drug administration and 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00, 48:00 h after drug administration
Population: The pharmacokinetic set (PKS) included all subjects in the treated set who provided at least one observation for at least one primary (PK) endpoint without important protocol violations relevant to the evaluation of PK and no vomiting must have occurred at or before two times the median tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Deleobuvir Trial Formulation II: Trial formulation II film-coated tablets.
  600 mg Deleobuvir (3 tablets à 200 mg). Oral administration with 240 mL water directly after a standard normal breakfast.
- Deleobuvir Final Formulation: Final formulation film-coated tablets.
  600 mg Deleobuvir (3 tablets à 200 mg). Oral administration with 240 mL water directly after a standard normal breakfast.
- Deleobuvir Final Formulation Modified: Final formulation modified film-coated tablets.
  600 mg Deleobuvir (3 tablets à 200 mg). Oral administration with 240 mL water directly after a standard normal breakfast.
Arm/Group | Deleobuvir Trial Formulation II | Deleobuvir Final Formulation | Deleobuvir Final Formulation Modified
Number analyzed (Participants) | 13 | 15 | 14
nmol*h/L | 10600 (45.0) | 12400 (57.3) | 13600 (66.0)
Statistical Analysis 1: Comparison: Deleobuvir Trial Formulation II vs Deleobuvir Final Formulation; Relative bioavailability comparison of Deleobuvir Trial Formulation II (reference) and Deleobuvir Final Formulation (test) in pairwise comparison. (reference : test); Test type: Superiority or Other; Ratio (%) = 123.4, 90% CI 2-sided [108.0 to 141.1], Standard Deviation 17.1 — The estimate of the relative bioavailability (%) is adjusted for the period effects in the ANOVA. The standard deviation is actually the gCV. CIs are based on the residual error from ANOVA, considering only the data from the 2 compared treatments
Statistical Analysis 2: Comparison: Deleobuvir Final Formulation vs Deleobuvir Final Formulation Modified; relative bioavailability comparison of Deleobuvir Final Formulation modified (test) and Deleobuvir Final Formulation (reference) in pairwise comparison. (reference : test); Test type: Superiority or Other; Ratio (%) = 109.8, 90% CI 2-sided [88.6 to 136.1], Standard Deviation 28.8 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Cmax
Description: Maximum measured concentration of Deleobuvir in plasma. The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: 1:00 h before drug administration and 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00, 48:00 h after drug administration
Population: The pharmacokinetic set (PKS).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Deleobuvir Trial Formulation II | Deleobuvir Final Formulation | Deleobuvir Final Formulation Modified
Number analyzed (Participants) | 13 | 15 | 14
nmol/L | 2460 (48.3) | 2990 (53.6) | 3070 (73.1)
Statistical Analysis 1: Comparison: Deleobuvir Trial Formulation II vs Deleobuvir Final Formulation; relative bioavailability comparison of Deleobuvir Final Formulation (test) and Deleobuvir Trial Formulation II (reference) in pairwise comparison. (test : reference); Test type: Superiority or Other; Ratio (%) = 122.5, 90% CI 2-sided [107.9 to 139.1], Standard Deviation 16.1 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Deleobuvir Final Formulation vs Deleobuvir Final Formulation Modified; relative bioavailability comparison of Deleobuvir Final Formulation modified (test) and Deleobuvir Final Formulation (reference) in pairwise comparison. (test : reference); Test type: Superiority or Other; Ratio (%) = 107.6, 90% CI 2-sided [83.1 to 139.4], Standard Deviation 35.0 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) occurring up to 2 days (48 h) after single intake of Deleobuvir tablets were assigned to the respective treatment period.
Description: The volunteers were required to report spontaneously any AEs (and time of onset, duration, intensity). In addition, each volunteer was assessed regularly by the medical staff throughout the clinical trial (including prior to discharge from the trial centre) as well as at the end of observation and whenever necessary as deemed by the investigator.
Groups:
- Deleobuvir (Total): All subjects while on treatment with Deleobuvir, i.e. there is no distinction between the 3 formulations.
Arm/Group | Deleobuvir Trial Formulation II | Deleobuvir Final Formulation | Deleobuvir Final Formulation Modified | Deleobuvir (Total)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/16 | 4/17 | 3/18 | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deleobuvir Trial Formulation II (N=16) | Deleobuvir Final Formulation (N=17) | Deleobuvir Final Formulation Modified (N=18) | Deleobuvir (Total) (N=18)
Headache (Nervous system disorders) | 3 | 4 | 2 | 5
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes